CLINICAL TRIAL: NCT05982613
Title: Effectiveness of Standard Therapy of Acne Vulgaris Based on Clinical Practice Guidelines (CPG) in Indonesia
Brief Title: Effectiveness of Standard Therapy of Acne Vulgaris
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: Department of Dermatology and Venereology, Faculty of Medicine Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia (Unknown); Ministry of Education, Culture, Research, and Technology of the Republic of Indonesia (Unknown)
Responsible Party: Principal Investigator, dr. Maria Clarissa Wiraputranto, Principal Investigator, Indonesia University
Other Study IDs: UIDV
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; clinical practice guideline; Indonesia; effectiveness; therapy
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General: This research is an observational study. There was no control and experimental group.

SUMMARY:
This study was to evaluate the effectiveness of standard therapy for acne vulgaris (AV) based on the clinical practice guidelines (CPG) in Indonesia. The main questions it aims to answer were:

1. How is the clinical characteristics of patients with AV in dr.Cipto Mangunkusumo Hospital?
2. How is the effectiveness of standard therapy for AV based on the CPG in Indonesia in reducing the number of non-inflammatory, inflammatory, and total lesions and degree of acne severity?

The clinical pratice guideline (CPG) used for analysis was CPG by dr.Cipto Mangunkusumo Hospital 2017 in line with the date of patient visit. Data of 724 patients with AV in dr.Cipto Mangunkusumo Hospital as recorded in the medical records were assessed for eligibility. Data of 3-month-follow-up data of included subjects were collected and analyzed.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of standard therapy for acne vulgaris (AV) based on the guidelines in Indonesia Design: An analytical retrospective observational study conducted from April 2023 through July 2023 using medical records of new acne patients between 2017 to 2019 from Dr. Cipto Mangunkusumo National Central General Hospital. A total sample of patients with AV who received standard therapy for acne vulgaris based on the guideline by Dr.Cipto Mangunkusumo Hospital in 2017 and not associated with systemic diseases or drugs were included. Patients were classified into mild, moderate, or severe acne using Lehmann grading system. Primary outcomes were changes in the number of non-inflammatory, inflammatory, and total lesions, and the proportion of acne severity after 3 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* New patients with acne vulgaris in the year 2017 to 2019
* Complete medical record data of 3-month follow-up, including data of: name, medical record number, sex, age, job, level of education, visit date, number of non-inflammatory, inflammatory, and total acne lesions, diagnosis of acne vulgaris based on Lehmann grading system
* Acne treatment based on clinical practice guideline by dr.Cipto Mangunkusumo Hospital 2017

Exclusion Criteria:

* Follow-up data less than 3 times in 3 months
* Incomplete medical record
* AV diagnosis without data on severity
* History of systemic diseases associated with acne such as polycystic ovarian syndrome and Cushing syndrome
* History of allergy with one or more standard acne therapy based on the clinical practice guideline
* Received acne therapy not aligned with clinical practice guideline by dr.Cipto Mangunkusumo Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New patients with acne vulgaris coming to the dermatology outpatient clinic in dr.Cipto Mangunkusumo hospital dated 2017 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change in non-inflammatory acne lesion count | week-12
  Change in the sum of the number of open and closed comedones
Change in inflammatory acne lesion count | week-12
  Change in the sum of the number of papules, pustules, nodes, and cysts
Change in total acne lesioncount | week-12
  Change in the sums of the number of non-inflammatory and inflammatory lesions
Change in acne severity | week-12
  Change in the acne severity based on Lehmann grading system (2002), which classified acne into mild, moderate, and severe

CONTACTS AND LOCATIONS:
Locations (1):
- dr.Cipto Mangunkusumo National Central General Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goh C, Cheng C, Agak G, et al. Acne vulgaris. In: Kang S, Amagai M, Bruckner AL, et al., eds. Fitzpatrick's Dermatology. 9th ed. McGraw-Hill; 2019:1391-1418.
- [Background] Wasitaatmadja SM, ed. Acne [Akne]. Badan Penerbit Fakultas Kedokteran Universitas Indonesia; 2018.
- [Background] Wasitaatmadja SM, Arimuko A, Norawati L, Bernadette I, Legiawati L, eds. Acne Management Guideline in Indonesia: Results Summary of Indonesian Acne Expert Meeting 2015 [ Pedoman Tata Laksana Akne Di Indonesia: Resume Hasil Indonesian Acne Expert Meeting 2015]. 2nd ed. Kelompok Studi Dermatologi Kosmetik Indonesia PERDOSKI; 2016.
- [Background] Tan AU, Schlosser BJ, Paller AS. A review of diagnosis and treatment of acne in adult female patients. Int J Womens Dermatol. 2017 Dec 23;4(2):56-71. doi: 10.1016/j.ijwd.2017.10.006. eCollection 2018 Jun. PMID 29872679
- [Background] Widaty S, Soebono H, Nilasari H, et al., eds. Akne. In: Clinical Practice Guidelines for Dermatology and Venereology Specialists in Indonesia [Panduan praktik klinis bagi dokter spesialis kulit dan kelamin di Indonesia]. Perhimpunan Dokter Spesialis Kulit dan Kelamin Indonesia (PERDOSKI); 2017:248-254.
- [Background] Department of Dermatology and Venereology dr. Cipto Mangunkusumo National Central General Hospital. Clinical Practice Guideline for Acne Vulgaris [Panduan Praktik Klinis Akne Vulgaris]. RSCM; 2017.
- [Background] Lehmann HP, Robinson KA, Andrews JS, Holloway V, Goodman SN. Acne therapy: a methodologic review. J Am Acad Dermatol. 2002 Aug;47(2):231-40. doi: 10.1067/mjd.2002.120912. PMID 12140469